CLINICAL TRIAL: NCT03959891
Title: Clinical Trial to Evaluate Safety and Anti-tumor Activity of AKT Inhibitor, Ipatasertib,With Endocrine Therapy With/Without CDK 4/6 Inhibitor for Patients With Metastatic Hormone Receptor Positive Breast Cancer (TAKTIC)
Brief Title: AKT Inhibitor, Ipatasertib, With Endocrine and CDK 4/6 Inhibitor for Patients With Metastatic Breast Cancer (TAKTIC)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Seth A. Wander, M.D., Ph.D., Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-086
Record Dates: First submitted 2019-05-15; First posted 2019-05-22 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ipatasertib; Fulvestrant; Aromatase Inhibitors; Letrozole; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fulvestrant + Ipatasertib (Experimental): * Ipatasertib will be administered orally on a daily basis
  * Fulvestrant would be administered as intra-muscular injection twice a month for the first cycle, and then monthly for all other cycles.
  Interventions: Drug: Ipatasertib; Drug: Fulvestrant
- Aromatase Inhibitor + Ipatasertib (Experimental): * Ipatasertib will be administered orally on a daily basis
  * Aromatase inhibitors will be administered orally on a daily basis
  Interventions: Drug: Ipatasertib; Drug: Aromatase Inhibitor
- Fulvestrant + Ipatasertib +Palbociclib (Experimental): * Ipatasertib will be administered orally on a 3 week on and 1 week off schedule
  * Fulvestrant would be administered as intra-muscular injection twice a month for the first cycle, and then monthly for all other cycles.
  * Palbociclib will be administered orally on a 3 week on and 1 week off schedule
  Interventions: Drug: Ipatasertib; Drug: Fulvestrant; Drug: Palbociclib

INTERVENTIONS:
Drug: Ipatasertib — Ipatasertib is a type of inhibitor that is believed to work by inhibiting Akt.
  Other Names: GDC-0068
Drug: Fulvestrant — Hormone therapies work by stopping the production of a certain hormone, blocking hormone receptors, or substituting chemically similar agents for the active hormone, which cannot be used by the tumor cell.
  Other Names: Falsodex
  Arms: Fulvestrant + Ipatasertib; Fulvestrant + Ipatasertib +Palbociclib
Drug: Aromatase Inhibitor — Letrozole is an aromatase inhibitor. This means it blocks the enzyme aromatase (found in the body's muscle, skin, breast and fat), which is used to convert androgens (hormones produced by the adrenal glands) into estrogen. In the absence of estrogen, tumors dependent on this hormone for growth will shrink.
  Other Names: Letrozole
  Arms: Aromatase Inhibitor + Ipatasertib
Drug: Palbociclib — Palbociclib (Ibrance®) is a drug that can be used along with an aromatase inhibitor to treat women with advanced hormone receptor-positive breast cancer. Palbociclib is a reversible small molecule cyclin-dependent kinase (CDK) inhibitor. The drug blocks proteins in the cell called cyclin-dependent kinase (CDK) 4 and CDK 6. In hormone positive breast cancer cells, blocking these proteins helps stop the cells from dividing to make new cells. It helps prevent the cells from moving from G1 to S cell cycle phase in the division process. This slows cancer growth.
  Other Names: Ibrance
  Arms: Fulvestrant + Ipatasertib +Palbociclib

SUMMARY:
This study is exploring the safety/tolerabtility and preliminary efficacy of the combination of Ipatasertib with Aromatase inhibitor or Fulvestrant for patients with metastatic HR+ breast cancer.

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational drug and also tries to define the appropriate dose of the investigational drug to use for further studies. "Investigational" means that the drug is being studied.

The U.S. Food and Drug Administration (FDA) has not approved ipatasertib as a treatment for any disease.

The FDA has approved fulvestrant, the aromatase inhibitors, and palbociclib as treatment options for this disease.

This research study will evaluate the safety and tolerability of ipatasertib in combination with an aromatase inhibitor or fulvestrant with or without palbociclib.

Resistance to standard of care treatment for people with your type of cancer is common. Stopping (inhibiting) an enzyme called Akt in the cancer cells may overcome resistance to the standard of care treatment. Ipatasertib is a type of inhibitor that is believed to work by inhibiting Akt. Through the different combinations of ipatasertib and the standard of care drugs, the chance of cancer cells becoming resistant to the standard of care drugs may decrease, causing the cancer cells to stop growing and spreading.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (≥ 18 years of age) with biopsy proven HR+/HER2 negative breast cancer; HR+ defined as ≥1% positivity for ER, and/or PR (≥1%), as per local assessment. HER2 as per standard CAP guidelines (local assessment).
* Postmenopausal women with locally advanced or metastatic BC. Patients must be postmenopausal women as defined by one of the following:

  * Women >60 years OR
  * Women ≤60 years, and any one of following:

    * LH and FSH level in the postmenopausal range according to institutional standards
    * s/p post bilateral surgical oophorectomy.
    * Premenopausal/perimenopausal women on gonadotropin-releasing hormone agonist (to be continued during study) and estradiol level in the postmenopausal range according to institutional standards
* Disease progression on at least one prior therapy for metastatic disease, including endocrine therapy with/without CDK 4/6 inhibitor (palbociclib or ribociclib or abemaciclib). Disease recurrence during/within 12 month of (neo)adjuvant endocrine therapy (with/without CDK 4/6 inhibitor) will count as one prior therapy for this definition.
* ECOG Performance Status 0 - 2
* Left ventricular ejection fraction (LVEF) ≥ 50%
* Evaluable or measurable disease: at least one lesion that can be accurately measured in at least one dimension ≥ 20 mm with conventional imaging techniques or ≥ 10 mm with spiral CT or MRI. Bone lesions in the absence of measurable disease as defined above is also acceptable.
* Discontinuation of prior breast cancer therapies, including endocrine therapy, for 14 days (non-myelosuppressive) or 21 days (myelosuppressive). Wash-out for Fulvestrant and tamoxifen will be 28 days.
* Prior mTOR inhibitor and/or PI3K inhibitor allowed (all arms)
* Prior aromatase inhibitor is allowed (all arms)
* Adequate bone marrow function: ANC ≥ 1000/mm3, hemoglobin ≥9 g/dl, and platelets ≥ 100,000/mm3.
* Adequate hepatic function: Total bilirubin < 1.5mg/dL, AST and ALT < 3X Institutional ULN (or 5 X Institutional ULN in presence of hepatic mets).
* Adequate renal function: Calculated creatinine clearance ≥ 30 mL/min
* Fasting blood glucose <140 mg/dL, and hemoglobin A1c <7.
* Signed informed consent and agree to comply with study procedures.

Exclusion Criteria:

* Participants with progressive CNS metastatic disease. Patients with stable CNS metastasis would be eligible, provided mets radiologically stable for atleast one month, and patient is not actively taking steroids.
* Participants who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Prior use of AKT inhibitor (any setting)
* Treatment with strong CYP3A inhibitors or strong CYP3A inducers within 14 days or 5 drug-elimination half-lives, whichever is longer, prior to initiation of study treatment. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list such as http://medicine.iupui.edu/clinpharm/ddis/table.aspx; medical reference texts such as the Physicians' Desk Reference may also provide this information. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product.
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., inflammatory bowel disease, ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality including any of the following:

  * History of angina pectoris, symptomatic pericarditis, coronary artery bypass graft (CABG) or myocardial infarction within 6 months prior to study entry.
  * Documented cardiomyopathy.
  * History of cardiac failure, significant/symptomatic bradycardia, Long QT syndrome, family history of idiopathic sudden death or congenital long QT syndrome or any of the following:
  * Known risk to prolong the QT interval or induce Torsade's de Pointes.
  * Uncorrected hypomagnesemia or hypokalemia.
  * Systolic Blood Pressure (SBP) >160 mmHg or <90 mmHg.
  * Bradycardia (heart rate <50 at rest), by ECG or pulse.
  * On screening, inability to determine the QTcF interval on the ECG (i.e.: unreadable or not interpretable) or QTcF >450 screening ECG (based on a mean of 3 ECGs).
* HIV-positive participants on combination antiretroviral therapy are ineligible. These participants are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* History of Type I or Type II diabetes mellitus requiring insulin. Patients who are on a stable dose of oral diabetes medication ≥ 2 weeks prior to initiation of study treatment are eligible for enrollment. Patients must meet the laboratory eligibility criteria for fasting blood glucose and hemoglobin A1c as outlined in the inclusion criteria.
* Pregnant women are excluded from this study because the safety of study medications is not established in pregnant women.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception throughout the study and for 8 weeks after study drug discontinuation. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of bilateral oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential. Highly effective contraception methods include:
* Total abstinence when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
* Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
* Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
* In case of use of oral contraception, women should have been stable on the same pill for a minimum of 3 months before taking study treatment. Note: While oral contraceptives are allowed, they should be used in conjunction with a barrier method of contraception due to unknown effect of drug-drug interaction.
* For Arm A only: patients who have received prior fulvestrant.
* For Arm C only: h/o of intolerable toxicity to CDK 4/6 inhibitor resulting in treatment discontinuation due to toxicity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2022-12-25 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 2 years
  grade 1-5 (CTCAE)

SECONDARY OUTCOMES:
Progression Free Survival | 2 years
  Kaplan-Meier Analysis
Overall Response Rate | 2 years
  RECIST criteria
Complete Response | 2 Years
  RECIST criteria
Partial Response | 2 years
  RECIST criteria
Overall Survival | 2 Years
  Kaplan-Meier Analysis

CONTACTS AND LOCATIONS:
Overall Officials: Seth Wander, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BCH - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu MGH - Contact the Partners Innovations team at http://www.partners.org/innovation